CLINICAL TRIAL: NCT03013829
Title: Kidney Paired Donation: A Randomized Trial to Increase Knowledge and Informed Decision-Making
Brief Title: Kidney Paired Donation Video-Based Education Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); Erie County Medical Center (Other)
Responsible Party: Principal Investigator, James Rodrigue, Vice Chair of Clinical Research, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016P000409
Record Dates: First submitted 2016-12-29; First posted 2017-01-09 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Kidney Paired Donation
Keywords: Kidney Paired Donation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Potential LKDs and recipients will receive standard-of-care LD (Live Donor) and KPD education. As noted previously, during standard care, incompatible potential LKDs are informed of the KPD option and the potential LKD is provided with living donation information and a link to the UNOS KPD website, which includes a written description of KPD. This information is available in English and Spanish. For those who do not have internet access, the written educational materials are mailed. The potential LKD is advised to call the donor nurse coordinator with any questions about KPD and/or to initiate the full donation evaluation. This process occurs for the intended recipient only if their potential donor decides to initiate the full evaluation.
  For study purposes, potential LKDs and waitlisted recipients assigned to the UC group will be sent an email after randomization, which will include a link and a reminder to review their transplant center's standard of care educational materials.
- Video-Based KPD education (Experimental): LKDs and recipients assigned to the video-based KPD education group will receive the same living donation and KPD educational materials as those in the UC group. Also, as in the UC group, they will be encouraged by the site coordinator to review the educational materials. In addition, following randomization to this group, participants will be sent an email encouraging them to watch the embedded KPD education video. This video will be professionally designed and will highlight the operational features of KPD and address the specific barriers highlighted in our formative research. The primary goal of these sessions is to increase living donation and KPD knowledge of risks and benefits and to reduce specific concerns that are based on inaccurate information. The intent is not to persuade LKDs or recipients to pursue living donation or KPD, but to ensure that they have sufficient information to make an informed choice that is consistent with their own values and preferences.
  Interventions: Behavioral: KPD Educational Video

INTERVENTIONS:
Behavioral: KPD Educational Video — LKDs and recipients assigned to the video-based KPD education group will receive the same living donation and KPD educational materials as those in the UC group. Also, as in the UC group, they will be encouraged by the site coordinator to review the educational materials. In addition, following randomization to this group, participants will be sent an email encouraging them to watch an embedded KPD education video. This video will be professionally designed and will highlight the operational features of KPD and address the specific barriers highlighted in our formative research. The primary goal of these sessions is to increase living donation and KPD knowledge of risks and benefits and to reduce specific concerns that are based on inaccurate information. The intent is not to persuade LKDs or recipients to pursue living donation or KPD, but to ensure that they have sufficient information to make an informed choice that is consistent with their own values and preferences.
  Arms: Video-Based KPD education

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a targeted educational approach designed to increase knowledge about the risks and benefits of living donation generally and KPD (Kidney Paired Donation) specifically, enhance KPD self-efficacy, reduce KPD concerns, and facilitate informed decision-making about KPD among potential live kidney donor and kidney transplant patients.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (RCT) to examine the effectiveness of a video-based KPD education intervention to improve knowledge, self-efficacy, concerns, and informed decision-making about KPD among potential live kidney donor and kidney transplant patients.

There will be equal allocation of LKDs and intended recipients to both KPD education conditions: (1) Usual Care (UC) group and (2) UC plus video-based KPD education group. All enrolled LKDs and intended recipients will complete a baseline survey and another survey 2 weeks post-intervention. Additionally, follow-up data will be gathered on KPD decision-making, participation, and reasons for non-participation at 3 months post-intervention.

Settings and target population:

The study will be conducted at three kidney transplant programs in the United States: Beth Israel Deaconess Medical Center (BIDMC; Boston, MA), the Medical University of South Carolina (MUSC; Charleston, SC), and Erie County Medical Center (ECMC; Buffalo, NY). BIDMC will act as the coordinating center for this study and will be responsible for study design, oversite, reporting, updates, and final data analysis. MUSC and ECMC will rely on the CCI at BIDMC for review. This study will target potential LKDs and their intended recipients.

Randomization:

Random assignment to the usual education or usual education plus video intervention group will occur within the 48 hours following completion of the baseline survey. The BIDMC study coordinator will oversee randomization after receiving an automated notification of baseline completion by participants from all study sites. Randomization will be done with the LKD, with the randomized group matched to the intended recipient. We have decided to ensure that the randomized group is the same for any LKD-recipient pairs to reduce the risk of contamination, which is a critical threat to internal validity in this type of study. For instance, if a LKD was assigned to the KPD video-based education group and their intended recipient was assigned to the UC group, there is the real possibility that there would be some diffusion of treatments in which the LKD discusses some elements of the intervention with the recipient and this, in turn, may influence the recipient's living donation and KPD knowledge, concerns, and decision-making processes. A simple unrestricted random allocation sequence will be used. We will use REDCap to generate the randomization sequence, which will be accessible to the site coordinators and transplant educators. The PI and Co-Investigators will be blinded to the subjects' allocation assignment.

Interventions:

Usual Care (UC) Living Donation and KPD Education:

Potential LKDs and recipients will receive living donation and KPD-specific education as they usually do at their respective kidney transplant programs.

Typically, potential LKDs are informed of their incompatibility during a phone call with the donor nurse coordinator. At this time, the KPD option is described and the potential LKD is provided with kidney paired donation information. This information is available in English and Spanish. For those who do not have internet access, the written educational materials are mailed. The potential LKD is advised to call the donor nurse coordinator with any questions about KPD and/or to initiate the full donation evaluation. An identical KPD educational process occurs for the intended recipient, although this is done with their own transplant nurse coordinator and only if their potential donor decides to initiate the full donation evaluation.

For study purposes, we will approach waitlisted recipients and any potential donors who complete an online health screening. LKDs and recipients assigned to the UC group will be sent an email after randomization, which will include a reminder to visit the usual educational websites and link to the usual care brochures. Participants will only be shown the materials provided as standard of care at their respective institutions.

Video-Based KPD Education:

LKDs and recipients assigned to the video-based KPD education group will receive the same living donation and KPD educational materials as those in the UC group. Also, as in the UC group, they will be encouraged by the site coordinator to review the educational materials. In addition, following randomization to this group, participants will be sent an email encouraging them to watch the embedded KPD education video. This video will be professionally designed and will highlight the operational features of KPD and address the specific barriers highlighted in our formative research. The primary goal of these sessions is to increase living donation and KPD knowledge of risks and benefits and to reduce specific concerns that are based on inaccurate information. The intent is not to persuade LKDs or recipients to pursue living donation or KPD, but to ensure that they have sufficient information to make an informed choice that is consistent with their own values and preferences.

Assessment Time-points:

Study data will be collected from participants at three different time points.

Baseline. Participants will complete a 30-minute online assessment via REDCap following email consent but prior to randomization. The questionnaire assessment will gather sociodemographic information, assess primary and secondary outcomes, and measure important covariates.

Post-Intervention. Two weeks after randomization, participants will complete a 20-minute REDCap assessment of the primary and secondary outcomes, uptake of the written and video educational elements, any discussions they have had with others about living donation or KPD, educational intervention process and evaluation, and any steps they have taken to pursue further donation evaluation. The rationale for the timing of this assessment is to re-assess the primary and secondary outcomes in close proximity to the delivery of living donation and KPD-specific education yet that provides sufficient time for the participant to assimilate and consider the information acquired.

Follow-up. Three months following the living donation and KPD-specific education, participants will complete a final REDCap assessment on living donation and KPD knowledge, as well as a brief assessment to learn of their final decision regarding living donation and the factors that contributed to it. The rationale for the timing of this follow-up assessment is that the vast majority of incompatible potential LKDs and recipients who have been offered KPD have achieved a final disposition within this time period.

ELIGIBILITY:
Inclusion Criteria:

LKDs

* Speaks English or Spanish
* Completed the initial living donation health screening

Transplant Candidates

* Speaks English or Spanish
* On that transplant waitlist (active or inactive)

Exclusion Criteria:

LKD's

* Non-directed (i.e., anonymous) potential LKDs
* Previously undergone donor evaluation
* Participation in another study to increase knowledge about living donation/LDK

Transplant Candidates

* Had a prior LDKT
* Previously enrolled in a KPD program
* Previous or current participation in another study to increase knowledge about living donation/LDKT
* Listed for a liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Living Donation and KPD Knowledge | at baseline
  A questionnaire will be used to assess living donation and KPD knowledge.
Living Donation and KPD Knowledge | 2 weeks post-intervention
  A questionnaire will be used to assess living donation and KPD knowledge.
Living Donation and KPD Knowledge | three months post-intervention
  A questionnaire will be used to assess living donation and KPD knowledge.

SECONDARY OUTCOMES:
Living Donation and KPD Concerns | at baseline
  Living donation and KPD concerns will be assessed using a Concerns about Living Donation scale and the Kidney Exchange Concerns (KEC) questionnaire.Questionnaire results will be aggregated to evaluate concerns about living donation and KPD.
Living Donation and KPD Concerns | 2 weeks post-intervention
  Living donation and KPD concerns will be assessed using a Concerns about Living Donation scale and the Kidney Exchange Concerns (KEC) questionnaire. Questionnaire results will be aggregated to evaluate concerns about living donation and KPD.
Informed Decision-Making | at baseline
  The investigators will measure living donation and KPD informed decision-making using five true-false items.
Informed Decision-Making | 2 weeks post-intervention
  The investigators will measure living donation and KPD informed decision-making using five true-false items.
Living Donation and KPD Self-Efficacy | at baseline
  The investigators will assess self-efficacy using a measure developed for the current NIDDK (National Institute of Diabetes and Digestive and Kidney Diseases)-funded House Calls RCT. This measure includes a list of actions or behaviors that are related to KPD, to which participants will indicate their level of confidence in carrying them out.
Living Donation and KPD Self-Efficacy | 2 weeks post-intervention
  The investigators will assess self-efficacy using a measure developed for the current NIDDK (National Institute of Diabetes and Digestive and Kidney Diseases)-funded House Calls RCT. This measure includes a list of actions or behaviors that are related to KPD, to which participants will indicate their level of confidence in carrying them out.
Living Donation and KPD Discussions | at baseline
  For the House Calls RCT, the investigators developed and validated a measure designed to assess the amount of time individuals spend talking to others about living donation. This measure asks whether the LKD or intended recipient talked to the donor/recipient, family members, friends, or healthcare providers about living donation and KPD, and if so, approximately how much time was spent discussing donation (TALKeD).
Living Donation and KPD Discussions | 2 weeks post-intervention
  For the House Calls RCT, the investigators developed and validated a measure designed to assess the amount of time individuals spend talking to others about living donation. This measure asks whether the LKD or intended recipient talked to the donor/recipient, family members, friends, or healthcare providers about living donation and KPD, and if so, approximately how much time was spent discussing donation (TALKeD).

OTHER OUTCOMES:
Living donation and KPD Activation- Evaluation of Actions Taken | three months post-intervention
  As part of the final follow-up assessment, the investigators will assess living donation and KPD activation, which asks participants to indicate whether they spoke to the donor/recipient about living donation and KPD, pursued further evaluation for living donation and KPD, entered the KPD registry, and/or donated or received a transplant. Participants will also be asked about reasons for not pursuing further evaluation or not registering for KPD. This outcome will measure action steps taken with regards to living donation and KPD.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Erie County Medical Center, Buffalo, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No